CLINICAL TRIAL: NCT06763536
Title: Testing Oral Nicotine Pouches to Reduce Smoking-Related Cancer in Rural Appalachia
Brief Title: Oral Nicotine Pouches Versus Nicotine Replacement Therapy to Reduce Cigarette Use for Smokers in Rural Appalachia
Acronym: ARISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brittney Keller-Hamilton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024C0064; NCI-2024-09181 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA289551-01 (NIH)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Carbon Monoxide; Tobacco Use Cessation Devices; albumin Rugby Park; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (oral nicotine pouch) (Experimental): SAMPLING PHASE: Participants receive 2 concentrations of three different flavors of oral nicotine pouches. Participants use the products ad libitum, starting with the lowest concentration, to determine their preferred concentration and flavor, over 2 weeks.
  SWITCH PHASE: Participants receive their preferred oral nicotine pouches and use them in place of cigarettes for 12 weeks.
  Participants complete surveys and have their carbon monoxide levels measured at various points throughout the study.
  OBSERVATION PHASE: After completion of the intervention, participants complete a final follow-up survey, along with a carbon monoxide measure, 14 weeks after the intervention ends.
  Interventions: Other: Carbon Monoxide Measurement; Other: Oral Nicotine Pouch; Other: Survey Administration; Other: Check-in Phone Calls
- Arm II (nicotine replacement therapy) (Active Comparator): SAMPLING PHASE: Participants receive 2 different strengths of nicotine replacement therapy patches and 2 different strengths and 3 different flavors of nicotine replacement therapy lozenges. Participants use the products ad libitum, starting with the lowest concentration, to determine their preferred concentration and flavor, over 2 weeks.
  SWITCH PHASE: Participants receive their preferred nicotine patches and lozenges and use them in place of cigarettes for 12 weeks.
  Participants complete surveys and have their carbon monoxide levels measured at various points throughout the study.
  OBSERVATION PHASE: After completion of intervention, participants complete a final follow-up survey, along with a carbon monoxide measure, 14 weeks after the intervention ends.
  Interventions: Other: Carbon Monoxide Measurement; Other: Nicotine Lozenge; Other: Nicotine Patch; Other: Survey Administration; Other: Check-in Phone Calls

INTERVENTIONS:
Other: Carbon Monoxide Measurement — Undergo carbon monoxide measurement
  Other Names: Carbon Monoxide; Covita iCOquit
Other: Nicotine Lozenge — Use nicotine lozenge
  Other Names: Rugby; Nicotine Replacement Therapy
  Arms: Arm II (nicotine replacement therapy)
Other: Oral Nicotine Pouch — Use oral nicotine pouch
  Other Names: ZYN
  Arms: Arm I (oral nicotine pouch)
Other: Nicotine Patch — Use nicotine patch
  Other Names: Rugby; Nicotine Skin Patch; Nicotine Transdermal Patch; Nicotine Replacement Therapy
  Arms: Arm II (nicotine replacement therapy)
Other: Survey Administration — measurements; data gathering
Other: Check-in Phone Calls — Check-in phone calls to study participants

SUMMARY:
This clinical trial compares the use of oral nicotine pouches to nicotine replacement therapy, consisting of nicotine patches and lozenges, to reduce cigarette use in smokers living in rural Appalachia. The lung and oral cancers that plague Appalachia are fueled by cigarette smoking. Oral nicotine pouches which contain nicotine but no tobacco leaf, present a new opportunity to reduce cancer risk among Appalachian adults who smoke. Oral nicotine pouches and nicotine replacement therapy may work well to reduce cigarette use for smokers in rural Appalachia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate short-term changes in cigarette smoking patterns, including switching, abstinence from cigarettes, and frequency of smoking between oral nicotine patches (ONPs) and NRT.

II. Compare product appeal, craving, withdrawal relief, and perceived cigarette dependence between ONPs and NRT.

III. Examine sustained changes in tobacco use behaviors, including abstinence from cigarettes, purchase of ONPs/NRT, and continued use of ONPs/NRT.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I:

SAMPLING PHASE: Participants receive 2 concentrations of three different flavors of oral nicotine pouches. Participants use the products ad libitum, starting with the lowest concentration, to determine their preferred concentration and flavor, over 2 weeks.

SWITCH PHASE: Participants receive their preferred oral nicotine pouches and use them in place of cigarettes for 12 weeks.

Participants complete surveys and have their carbon monoxide levels measured at various points throughout the study.

OBSERVATION PHASE: After completion of the intervention, participants complete a final follow-up survey, along with a carbon monoxide measure, 14 weeks after the intervention ends.

ARM II:

SAMPLING PHASE: Participants receive 2 different strengths of nicotine replacement therapy patches and 2 different strengths and 3 different flavors of nicotine replacement therapy lozenges. Participants use the products ad libitum, starting with the lowest concentration, to determine their preferred concentration and flavor, over 2 weeks.

SWITCH PHASE: Participants receive their preferred nicotine patches and lozenges and use them in place of cigarettes for 12 weeks.

Participants complete surveys and have their carbon monoxide levels measured at various points throughout the study.

OBSERVATION PHASE: After completion of intervention, participants complete a final follow-up survey, along with a carbon monoxide measure, 14 weeks after the intervention ends.

ELIGIBILITY:
Inclusion Criteria:

* Read and speak English
* 21 years or older
* Smoke ≥ 5 cigarettes per day for the past year
* Willing to use Oral Nicotine Pouches (ONP) or Nicotine Replacement Therapy (NRT)
* Live in a rural Appalachian County
* Have a smartphone and/or willing to use a smartphone for study purposes (smartphones may be provided to participants for study purposes only)
* Willing to blow air into a handheld study device
* If capable of becoming pregnant, verbal confirmation of not being pregnant based on urine pregnancy test results

Exclusion Criteria:

* Report currently using smoking cessation medications, NRT, or actively seeking treatment for smoking cessation
* Use of ONPs in past 3 months
* Use of Nicotine Replacement Therapies in past 3 months
* Use of other tobacco products > 10 days/month
* Unstable or significant medical condition
* Unstable or significant psychiatric conditions (past and stable conditions will be allowed)
* History of cardiac event or distress within the past 3 months
* Live in same household as another study participant.
* Currently pregnant, planning to become pregnant within 6 months, or breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemically verified 7-day point prevalence abstinence from cigarettes | At the end of the 12- week switch phase
  Statistical analyses will be performed using SAS 9.4. P-values less than 0.05 will be considered statistically significant. Will be presented as frequencies and proportions and compared with chi-squared tests.
Complete switching rate (Aim 1) | At the end of the 12-week switch phase
  Will be compared between arms using logistic regression analysis, adjusting for baseline variables as needed.
Abstinence from cigarettes (Aim 1) | At the end of the 12-week switch phase
  Will be compared between arms using logistic regression analysis, adjusting for baseline variables as needed.
Cigarettes smoked per day (Aim 1) | At the end of the 12-week switch phase
  If needed, will apply a normalizing transformation to the number of cigarettes smoked per day (e.g., taking the logarithm) before proceeding with the analysis as a means of removing the effects of potential outliers. Will compare cigarettes smoked per day between the two arms using linear regression analysis. The model will adjust for cigarettes smoked per day at baseline and other baseline variables if they are imbalanced.
Differences in product appeal (Aim 2) | From baseline to the end of the 12 week switch phase
  Will be adjusted for potential confounders including baseline variables such as age, gender, number of cigarettes smoked per day, and/or randomization stratification factors as necessary; normalizing transformations will be employed if needed.
Cigarette craving (Aim 2) | Up to the end of the 12 week switch phase
  Will be evaluated with linear regression models adjusting for appropriate confounders.
Withdrawal symptoms (Aim 2) | Up to the end of the 12 week switch phase
  Will be evaluated with linear regression models adjusting for appropriate confounders.
Change in nicotine dependence among participants who completely switched to their assigned study product (Aim 2) | From baseline to the end of the 12 weeks switch phase
  Using linear regression analysis, adjusting for baseline nicotine dependence.
Abstinence from cigarettes (Aim 3) | Up to the end of the 14 week observation phase
  Will be compared between arms using logistic regression analysis and will be evaluated with a logistic regression model.
Number of days the study products are used (Aim 3) | Up to the end of the 14 week observation phase
  Linear regression analysis will be used to compare the number of days the products are used. A normalizing transformation will be employed if needed and appropriate baseline characteristics will be adjusted for.
Purchase and continued use of the study products (Aim 3) | Up to the end of the 14 week observation phase
  Will be compared between the arms with logistic regression analysis, adjusting for all appropriate confounders.

CONTACTS AND LOCATIONS:
Overall Officials: Brittney L Keller-Hamilton, PhD, MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Wermert A, Brasky TM, Newton AM, Hinton A, Curran H, Ferketich AK, Carpenter MJ, Shields PG, Tomko P, Wagener TL, Keller-Hamilton B. Testing oral nicotine pouches versus nicotine replacement therapy for cigarette harm reduction in Appalachia: The ARISE study protocol. PLoS One. 2025 Dec 23;20(12):e0338503. doi: 10.1371/journal.pone.0338503. eCollection 2025. PMID 41433314
- See also: The Jamesline — http://cancer.osu.edu